CLINICAL TRIAL: NCT03600012
Title: Investigating of Effects of Lower Extremities Cycling Functional Electrıcal Stimulation Training On Gait Parameters In Children With Diplegic Cerebral Palsy
Brief Title: Effects of Lower Extremities Cycling Functional Electrıcal Stimulation Training in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Turker, principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 14/119
Record Dates: First submitted 2018-06-03; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Cerebral Palsy; Diplegic Cerebral Palsy
Keywords: Diplegic Cerebral Palsy; Cycling With Functional Electrical Stimulation; Gait Analysis; Functional Strenght Training; Quality of Life; Qxygen Consumption
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): intervention group: Cycling Functional Electrical Stimulation & Physiotherapy
  Children in intervention group were taken in a therapy program withRT 300 SLSA FES system for cycling functional electrical stimulation training additionly to physiotherapy program including weight shifting, knee and hip strenging and gait training for 8 weeks, 3 sessions in a week and 45 min per session.
  Interventions: Other: Cycling Functional Electrical Stimulation; Other: Physiotherapy
- control group (Active Comparator): control group: Physiotherapy
  Children with cp in control group were taken physiotherapy program including weight shifting, knee and hip strenging and gait training for 8 weeks, 3 times in a week, 45 min per session.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Cycling Functional Electrical Stimulation
  Arms: intervention group
Other: Physiotherapy

SUMMARY:
The aim of this study was to investigate the effects of cycling functional electrical stimulation applied to the lower extremities of children with spastic diplegic cerebral palsy (CP) on the gait parameters and daily living activities.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a broadly-defined neurological disorder that encompasses brain injury or malformation in a child's brain that occurs before, during, or immediately after birth and results in impaired motor control. Because of the broad definition of CP, people with CP can exhibit a very wide range of symptoms, and no two people with CP will exhibit the same symptoms. However, people with CP generally have difficulty moving parts of their bodies normally because of muscle weakness or paralysis, impaired muscle coordination, and/or spasticity. Impaired motor control can also be accompanied by intellectual impairment, seizures, or sensory impairment.

Physical impairment can severely limit participation in physical activity by people with CP, as is true for anyone with physical impairments. Lack of physical activity can lead to the development of any number of chronic diseases, especially in children with disabilities like CP. Exercise is an effective method for mitigating the negative secondary health effects of neuromuscular diseases like CP, but how can someone with CP exercise despite their impaired motor control, especially when 31% of children with CP have limited walking ability.

Cycling is an exercise that challenges the muscular and cardiovascular systems, potentially leading to improved health, fitness, and well-being. Cycling with functional electrical stimulation (FES) has been primarily used by people with spinal cord injury; improvements have been seen in bone mineral density, muscle strength (force-generating capacity), and cardiorespiratory measures. Recent reports indicated benefits for people after stroke; improvements in strength and motor control were seen when an FES cycling program was added to traditional rehabilitation. However, there have been no reports of FES cycling for children with CP.

Cycling with FES may be a suitable intervention for with CP because the seated position decreases balance demands, and FES can create or augment pedaling forces. Many people with CP may be incapable of generating sufficient forces during cycling to reach the exercise intensity needed for optimal fitness-related outcomes and musculoskeletal benefits.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy
* classified in levels I - II of the Gross Motor Function Classification System (GMFCS)
* able to follow and accept verbal instruction

Exclusion Criteria:

* any orthopaedic surgery or botulinum toxin injection in the past 6 months,
* children whose parents refused to participate

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Gait was assessed using a three-dimensional Gait Analysis motion system. | change from baseline gross motor funciton at 8 weeks
  Gait was assessed using a three-dimensional, seven-camera, VICON 512 motion measurement system (Oxford Metrics Ltd., Oxford, UK). The VICON Clinical Manager software was used for calculating and plotting temperospatial parameters, sagittal plane joint motion data, and kinematic data. Fifteen reflective markers were placed on specific anatomic landmarks bilaterally of the subject's pelvis, thighs, shanks and feet according to the marker protocol of Davis et al.
Walking energy expenditure measurements were done with breath by breath method. | change from baseline gross motor funciton at 8 weeks
  Walking energy expenditure measurements were done with breath by breath method using an open-circuit indirect calorimeter (Vmax 29c, Sensormedics, USA).

SECONDARY OUTCOMES:
Gross motor function was measured using GMFM. | change from baseline gross motor funciton at 8 weeks
  The GMFM measures capability, or what a child 'can do' in a standardized environment. Items include tasks related to lying and rolling, sitting, crawling and kneeling, standing, walking, running and jumping, with the most difficult items on the scale representing abilities obtained by children developing typically by 5 years of age. Each item is scored by observation on a four-point ordinal scale (0-3).
Modified Ashworth (MAS) scale was used to evaluate muscle tone. | change from baseline gross motor funciton at 8 weeks
  The MAS is a 6-point rating scale which assesses muscle tone by manually manipulating the joint through its available range of motion and clinically recording the resistance to passive movements.
The 30s Repetition Maximum test was used to assess functional muscle strength of the lower extremities. | change from baseline gross motor funciton at 8 weeks
  The three closed kinetic chain exercises of lateral step-up test, sit to stand, and attain stand through half knee were used.
Balance was assessed with pediatric balance scale (PBS). | change from baseline gross motor funciton at 8 weeks
  Functional balance was assessed using the PBS, which consists of 14 tasks similar to activities of daily living. The items are scored on a five-point scale (0, 1, 2, 3 or 4), with zero denoting an inability to perform the activity without assistance and four denoting the ability to perform the task with complete independence. The score is based on the time for which a position can be maintained, the distance to which the upper limb is capable of reaching in front of the body, and the time needed to complete the task. The maximum score is 56 points.
Dynamic balance was assessed withTime up & go test (TUG). | change from baseline gross motor funciton at 8 weeks
  TUG test a performance measure of speed to complete a sequenced functional mobility task. The TUG test measures, the time required for an individual to stand up from a standard chair with armrest, walk 3m, turn around, walk back to the chair, and sit down again. The test has been widely used in clinical practice as an outcome measure to evaluate functional mobility.
Daily living activity was assessed with Pediatric Evaluation of Disability Inventory. | change from baseline gross motor funciton at 8 weeks
  Pediatric Evaluation of Disability Inventory quantitatively measures functional performance. This questionnaire was administered in interview form to one of the child's caregivers who was knowledgeable about the performance of the child in typical activities and tasks of daily routine. The first part of the questionnaire was used. This assesses skills in the child's repertoire grouped into three functional categories: self-care (73 items), mobility (59 items) and social function (65 items). An item is scored 0 (zero) when the child is unable to perform the activity or 1 (one) when the activity is part of the child's repertoire of skills. The scores are totaled per category.
Quality of life was assessed withThe Child Health Questionnaire (CHQ-PF50). | change from baseline gross motor funciton at 8 weeks
  CHQ is a multidimensional generic health status questionnaire developed for clinicians and researchers interested in measuring children's functional health and well-being. It is available as a parent/proxy report for children aged 5-18 years and as a corresponding self-report for adolescents. The CHQ PF50 includes 13 single and multi-item scales that tap concepts contributing to overall functioning and well-being for children in the context of their family and social environments. One of the purported advantages of the CHQ PF50 is the availability of two summary scores (psychosocial and physical), which may be used in the evaluation of outcomes when information at the scale level is not practical.

CONTACTS AND LOCATIONS:
Overall Officials: yavuz yakut, prof.dr, Study Chair — Hacettepe University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerr C, McDowell B, McDonough S. Electrical stimulation in cerebral palsy: a review of effects on strength and motor function. Dev Med Child Neurol. 2004 Mar;46(3):205-13. doi: 10.1017/s0012162204000349. No abstract available. PMID 14995090
- [Background] Chiu HC, Ada L. Effect of functional electrical stimulation on activity in children with cerebral palsy: a systematic review. Pediatr Phys Ther. 2014 Fall;26(3):283-8. doi: 10.1097/PEP.0000000000000045. PMID 24819681
- [Background] Dodd KJ, Taylor NF, Damiano DL. A systematic review of the effectiveness of strength-training programs for people with cerebral palsy. Arch Phys Med Rehabil. 2002 Aug;83(8):1157-64. doi: 10.1053/apmr.2002.34286. PMID 12161840
- [Background] Fowler EG, Knutson LM, Demuth SK, Siebert KL, Simms VD, Sugi MH, Souza RB, Karim R, Azen SP; Physical Therapy Clinical Research Network (PTClinResNet). Pediatric endurance and limb strengthening (PEDALS) for children with cerebral palsy using stationary cycling: a randomized controlled trial. Phys Ther. 2010 Mar;90(3):367-81. doi: 10.2522/ptj.20080364. Epub 2010 Jan 21. PMID 20093327
- [Background] Fowler EG, Knutson LM, DeMuth SK, Sugi M, Siebert K, Simms V, Azen SP, Winstein CJ. Pediatric endurance and limb strengthening for children with cerebral palsy (PEDALS)--a randomized controlled trial protocol for a stationary cycling intervention. BMC Pediatr. 2007 Mar 21;7:14. doi: 10.1186/1471-2431-7-14. PMID 17374171
- [Background] Williams H, Pountney T. Effects of a static bicycling programme on the functional ability of young people with cerebral palsy who are non-ambulant. Dev Med Child Neurol. 2007 Jul;49(7):522-7. doi: 10.1111/j.1469-8749.2007.00522.x. PMID 17593125
- [Background] Johnston TE, Wainwright SF. Cycling with functional electrical stimulation in an adult with spastic diplegic cerebral palsy. Phys Ther. 2011 Jun;91(6):970-82. doi: 10.2522/ptj.20100286. Epub 2011 Apr 28. PMID 21527385
- [Background] Trevisi E, Gualdi S, De Conti C, Salghetti A, Martinuzzi A, Pedrocchi A, Ferrante S. Cycling induced by functional electrical stimulation in children affected by cerebral palsy: case report. Eur J Phys Rehabil Med. 2012 Mar;48(1):135-45. Epub 2011 Apr 20. PMID 21508913